CLINICAL TRIAL: NCT02483923
Title: Analgesic Effect to Postoperative Pain After Mastectomy: Ultrasound-guided Serratus Anterior Plane Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4-2015-0363
Record Dates: First submitted 2015-06-18; First posted 2015-06-29 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Breast Cancer
Keywords: serratus anterior block; ultrasound; breast cancer; postoperative pain
MeSH Terms: conditions — Breast Neoplasms; Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group S (Experimental)
  Interventions: Drug: Ultrasound guided serratus anterior block with ropivacaine
- Group C (Placebo Comparator)
  Interventions: Drug: intravenous PCA only

INTERVENTIONS:
Drug: Ultrasound guided serratus anterior block with ropivacaine — After induction of anesthesia, patients take ultrasound guided serratus anterior plane block with 0.5ml/kg of ropivacaine 0.375%. 30minutes before the end of operation, intravenous patient controlled analgesia (Basal rate 0ml/hr, 0.5mcg/kg of fentanyl, lock-out time 10minutes) is connected to patient.
  Arms: Group S
Drug: intravenous PCA only — same dose of intravenous patient controlled analgesia (Basal rate 0ml/hr, 0.5mcg/kg of fentanyl, lock-out time 10minutes) is connected to patient only.
  Arms: Group C

SUMMARY:
Ultrasound guided serratus anterior plane block may decrease acute postoperative pain and consumption of opioid after mastectomy.

ELIGIBILITY:
Inclusion Criteria:

1. ASA 1~3
2. Age 20~80
3. Breast cancer patient twho are scheduled for elective mastectomy

Exclusion Criteria:

1. Allergy to local anesthetics or contraindication to use of ropivacaine
2. Pregnancy
3. Severe cardiovascular disease
4. Renal failure
5. Liver failure
6. Neurologic and psychologic disease
7. Chronic treatment with analgesics
8. Previous history of mastectomy or thoracic surgery.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-06-16 (Actual); Primary Completion 2016-02-28 (Actual); Study Completion 2016-02-28 (Actual)

PRIMARY OUTCOMES:
Total opioid consumption | within 24 hrs after mastectomy
  Assessing total opioid consumption (total number of bolus injection and total dose of fentanyl via intravenous patient controlled analgesia) within 24hours after operation finished.

SECONDARY OUTCOMES:
Postoperative pain scale (Numeric rating scale 0-10) at PACU | chang from 3,6,12,24 to 48hrs after operation end
Total intraoperative remifentanil consumption(mcg) | within 24 hrs after mastectomy
Additional analgesics requirements (dose/number) | within 24 hrs after mastectomy
incidence and intensity of postoperative nausea and vomiting(NRS:0-10) | within 24 hrs after mastectomy
Total hospital staying time | within 24 hrs after mastectomy

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea